CLINICAL TRIAL: NCT05268562
Title: Impact of Ketamine Versus Propofol for Anesthetic Induction on Acute Kidney Injury and Renal Biomarkers in Cardiac Surgery
Brief Title: Ketamine and Kidney Injury in Cardiac Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erica D. Wittwer, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-004327
Record Dates: First submitted 2022-02-08; First posted 2022-03-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery
Keywords: Cardiopulmonary bypass
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anesthesia induction with Ketamine (Active Comparator): Subjects will receive Ketamine to begin anesthesia for their cardiac surgery.
  Interventions: Drug: Ketamine
- Anesthesia induction with Propofol (Active Comparator): Subjects will receive Propofol to begin anesthesia for their cardiac surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — 1-2 mg/kg induction with additional medication administered as needed to achieve intubating conditions
  Arms: Anesthesia induction with Ketamine
Drug: Propofol — 0.5-1 mg/kg induction with additional medication administered as needed to achieve intubating conditions
  Arms: Anesthesia induction with Propofol

SUMMARY:
The purpose of this study is to investigate the affects of ketamine use for anesthesia at the beginning of heart surgery on kidneys compared to the use of propofol.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for cardiac surgery at the Mayo Clinic in Rochester, Minnesota.
* Scheduled to undergo complex cardiac surgery with the use of cardiopulmonary bypass. Complex cardiac surgery will be defined as surgery involving more than one heart valve, redo-sternotomy procedures, or combined valvular and coronary artery bypass graft procedures (aortic repair not excluded if meets other criteria).

Exclusion Criteria:

* Left or right ventricular assist device implantation or explantation.
* Procedures not requiring cardiopulmonary bypass.
* Active infection or sepsis requiring antimicrobial therapy and/or vasopressor therapy (treated endocarditis is not excluded).
* Severe hepatic disease resulting in ascites.
* Pre-operative significant renal dysfunction including a baseline creatinine equal to or greater than 2 mg/dL or requiring dialysis.
* Immunosuppressive medication use (including current IV or oral steroids use, use of anti-rejection medications for transplant within 1 month, or chemotherapy within 6 months).
* Immunodeficiency syndrome including HIV/AIDS, leukemia, and multiple myeloma

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | Immediately postop up to 10 days postoperatively
  The incidence of acute kidney injury in patients following cardiac surgery

SECONDARY OUTCOMES:
Vasopressor use | Immediately post induction up to 30 minute following induction
  Compare mean total vasopressor doses, in norepinephrine equivalents, between groups following induction as a surrogate for hemodynamic differences

CONTACTS AND LOCATIONS:
Overall Officials: Erica D Wittwer, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials